CLINICAL TRIAL: NCT01771497
Title: Koning Breast CT (KBCT)-Guided Neoadjuvant Treatment of Breast Cancer Monitoring Phase I Trial
Brief Title: Koning Breast Computed Tomography Guided Neoadjuvant Treatment Monitoring
Status: Completed | Type: Observational
Sponsor: Koning Corporation (Industry)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: KBCT-005
Record Dates: First submitted 2012-12-13; First posted 2013-01-18 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2015-03

CONDITIONS: Breast Cancer
Keywords: Breast CT
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Women undergoing neoadjuvant therapy
  Interventions: Device: Koning Breast CT

INTERVENTIONS:
Device: Koning Breast CT — Koning Breast CT scans will be assessed at the beginning, mid-point and end of therapy.
  Other Names: Dedicated breast CT

SUMMARY:
The hypothesis of this study is that using Koning Breast CT during the neoadjuvant treatment of breast cancer will allow for accurate tumor localization and tumor volume measurement, leading to improved surgical and radiation therapy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age 18 years or older
* Any ethnicity
* Are undergoing neoadjuvant therapy for locally advanced breast cancer with either chemotherapy or hormonal therapy
* Is able to provide informed consent.

Exclusion Criteria:

* Pregnancy
* Lactation
* Women who are unable or unwilling to understand or to provide informed consent
* Women with physical limitations that may prohibit resting prone on the exam table, such as, but not limited to: frozen shoulder, recent heart surgery, pace maker.
* Women who are unable to tolerate study constraints.
* Women who have received radiation treatments to the thorax for malignant and nonmalignant conditions, such as (but not limited to):
* Treatment for enlarged thymus gland as an infant
* Irradiation for benign breast conditions, including breast inflammation after giving birth
* Treatment for Hodgkin's disease
* Women who have participated in a prior breast clinical trial that gave additional radiation dose, such as an additional mammogram.
* Women who have received large numbers of diagnostic x-ray examinations for monitoring of disease such as (but not limited to):
* Tuberculosis
* Severe scoliosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twelve female patients at least 18 years of age undergoing neoadjuvant therapy for locally advanced breast cancer with either chemotherapy or hormonal therapy will be recruited for this study. Inclusion of those patients 18 years or older is important since as it is the younger patients who present with breast cancer that often end up receiving neoadjuvant treatment.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2010-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Tumor volume change from baseline during neoadjuvant treatment | Baseline, mid-point (~3 months), and end of therapy (4-6 months)
  Tumor volume will be measured with KBCT imaging at the beginning of the therapy (baseline), mid-point of the therapy (about 3 months after the treatment starts) and end of therapy (about 4-6 months after the treatment starts). The volume change from the baseline during the treatment will be recorded.
  Adverse Events will be recorded as a measure of safety.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center Highland Breast Imaging Center, Rochester, New York, United States